CLINICAL TRIAL: NCT00616850
Title: Treatment of Postoperative Pain After Total Knee Arthroplasty Using Intravenous Lidocaine Infusion in Combination With Patient Controlled Analgesia Versus Continuous Femoral Block Catheter in Combination With Patient Controlled Analgesia: A Prospective, Randomized, Double-Blinded, Placebo-Controlled Study.
Brief Title: Treatment of Postoperative Pain After Total Knee Arthroplasy Using Intravenous Lidocaine Infusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Orthopedic surgeon that does our knee surgeries moved to a different location
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 57175
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Intravenous Lidocaine Infusion; Femoral Block Catheter
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Group A subjects will receive a continuous femoral block catheter and a Patient Controlled Analgesia (PCA).
  Interventions: Procedure: Continuous femoral catheter block
- Group B (Experimental): Group B subjects will receive a low dose lidocaine (1.33 mg/kg/hr) infusion and a Patient Controlled Analgesia.
  Interventions: Drug: Lidocaine
- Group C (Placebo Comparator): Group C subjects will receive placebo (preservative free normal saline) infusion and a Patient Controlled Analgesia.
  Interventions: Other: Preservative free normal saline

INTERVENTIONS:
Procedure: Continuous femoral catheter block — A constant infusion of ropivacaine 0.2% without epinephrine will be given to each subject via continuous femoral catheter in Group A.
  Arms: Group A
Drug: Lidocaine — Lidocaine 1.33mg/kg/hr continuous IV infusion following induction of general anesthesia to 24 hours postoperatively.
  Arms: Group B
Other: Preservative free normal saline — Preservative free normal saline 1.33mg/kg/hr continuous IV infusion following induction of general anesthesia to 24 hours postoperatively.
  Arms: Group C

SUMMARY:
Total knee replacement is often associated with severe postoperative pain, especially in the first 24 hours. Patient controlled analgesia (PCA) and continuous femoral block with PCA are commonly used to treat postoperative pain after total knee arthroplasty. However, PCAs use opioids. Opioids are excellent painkillers but their use is hampered by side effects such as nausea, vomiting, bowel dysfunction, urinary retention, pruritus, sedation and respiratory depression. We propose to test the hypothesis that adding a low dose lidocaine infusion to PCAs will lower the amount of opioids that these patients receive, thereby improving patient safety while still providing adequate analgesia. In addition, continuous femoral block has been shown to provide superior postoperative pain control when compared to morphine PCA. Therefore, postoperative pain levels of study subjects will be compared to those subjects who receive a combination of a continuous femoral block catheter with a PCA.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing a total knee arthroplasty
2. Be American Society of Anesthesiologist physical status 1,2, or 3
3. Be willing and capable of providing informed consent
4. Be English speaking

Exclusion Criteria:

1. Age greater than 80 years old or younger than 18 years old
2. Congestive hear failure
3. Hepatic insufficiency
4. Neurological disorders
5. Psychiatric disorders
6. Steroid treatment
7. History of atrial fibrillation
8. Chronic pain disorder with opioid treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Total PCA opioid consumption | 72 hours

SECONDARY OUTCOMES:
Time to first flatus | 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Schlunt, M.D., Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States